CLINICAL TRIAL: NCT04592926
Title: The Impact of Pre-Insertion Ultrasound for Lateral-Position Spinal in Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Pre-Insertion Ultrasound for Lateral-Position Spinal in Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Naida Margaret Cole, Staff Anesthesiologist, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020P
Record Dates: First submitted 2020-09-28; First posted 2020-10-19 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Cesarean Section; Spinal Anesthesia; Lumbar Ultrasound
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and observer who collects the outcome data will be blinded to group allocation. The anesthesiologist caring for the patient and the resident/fellow performing the spinal anesthetic will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Accuro ultrasound (Experimental)
  Interventions: Device: Accuro SpineNav3D
- Control (Sham Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Device: Accuro SpineNav3D — The intervention will consist of a pre-procedural scan of the lumbar spine using the handheld image guidance device, Accuro, to determine spinal landmarks and anticipated depth of the intrathecal space.
  Other Names: Accuro
  Arms: Accuro ultrasound
Other: Sham — The sham group will receive a pre-procedure sham scan (the handheld image guidance Accuro device will be placed on the back, but it will be turned off) followed by sham marking on the subject's back.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the impact of lumbar ultrasound anatomic mapping using the Accuro device on the number of needle redirections, when performing spinal anesthesia in the lateral decubitus position on patients undergoing elective cesarean delivery.

DETAILED DESCRIPTION:
Training in neuraxial placement most commonly occurs with patients in the sitting position, since it is easy to master. However lateral placement may be preferred in emergent situations and for patient comfort. In order to provide safe and effective anesthesia to parturients, providers must be competent with the technique in both sitting and lateral positions.

Ultrasound examination prior to spinal placement is a safe, non-invasive method of determining depth, midline, and interspinous location. Its use may decrease the number of needle insertions and needle passes in parturients in the sitting position, however little is known about the benefit of ultrasound use in the placement of lateral spinals.

The use of lumbar ultrasound with Accuro may improve success rates, safety, and the education of residents as they learn neuraxial placement in the lateral position. This will be the first study to examine the use of Accuro for lateral neuraxial placement.

The study investigators hypothesize that lumbar ultrasound with the handheld Accuro device by an experienced provider prior to spinal insertion will result in fewer needle redirections compared to palpation of landmarks when performed by anesthesia residents or fellows.

The two arms of the study are as follows:

Group 1: Control Group: sham pre-puncture ultrasound procedure with the handheld Accuro device turned off, followed by a sham marking on the participant's back using the Accuro locator marker attached to the device.

Group 2: Ultrasound Group: pre-puncture ultrasound with Accuro followed by marking placed at the L3-4 interspace in the midline using the attached Accuro locator marker.

All ultrasound exams will be performed by an unblinded physician study investigator.

All study participants will have a spinal anesthetic in lateral position performed by one of the residents or fellows participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* 18 years or older
* singleton pregnancy
* at least 37 weeks gestational age
* American Society of Anesthesiologists (ASA) Classification II
* body mass index (BMI) <35 kg/m2
* plan for elective and scheduled cesarean section with spinal anesthesia

Exclusion Criteria:

* patient refusal of spinal anesthesia
* uncorrected coagulopathy
* infection at the skin site of spinal placement
* increased intracranial pressure
* untreated hemodynamic instability
* history of scoliosis or spine surgery
* BMI >/=35 kg/m2
* allergy to local anesthetic
* allergy to opioids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Needle Redirections | through study completion, average of 3 hours
  Number of times the angle of the spinal introducer needle is adjusted, without exiting and re-entering the skin

SECONDARY OUTCOMES:
Number of Needle Passes | through study completion, average of 3 hours
  Number of times the spinal introducer needle exits the skin and re-enters the skin at a new location
Procedural Time | through study completion, average of 3 hours
  The time from subcutaneous injection of local anesthetic prior to spinal placement until the return of cerebrospinal fluid through the spinal needle is confirmed
Patient Satisfaction with procedure | through study completion, average of 3 hours
  Patient's rating of their satisfaction with the spinal procedure using a 0-10 numeric rating scale, as measured by a blinded study investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no current IPD sharing plan for this data.